CLINICAL TRIAL: NCT04924803
Title: Community Developed Technology-Based Messaging to Increase SARS-CoV-2 Vaccine Uptake Among People Who Inject Drugs
Brief Title: Community Developed Technology-Based Messaging to Increase COVID-19 Vaccine Uptake Among People Who Inject Drugs
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NDRI-USA, Inc. (Other)
Collaborators: New York Harm Reduction Educators (Unknown); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: COVID Vaccination; R01DA054990 (NIH)
Record Dates: First submitted 2021-06-09; First posted 2021-06-14 (Actual); Last update posted 2025-03-21 (Actual); Status verified 2025-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No video condition (Experimental): Participants in the no video condition will receive weekly text messages designed to increase vaccination among our sample.
  Interventions: Behavioral: No video
- Video text condition (Experimental): Participants in the video text condition will receive the text messages designed to increase vaccination among our sample, along with links to iteratively developed intervention videos
  Interventions: Behavioral: Video Text

INTERVENTIONS:
Behavioral: No video — Weekly text messages
  Arms: No video condition
Behavioral: Video Text — Weekly text messages including links to intervention videos
  Arms: Video text condition

SUMMARY:
People who inject drugs (PWID) experience disproportionate risk of being infected with SARS-CoV-2, the virus that causes COVID-19, yet due to stigma, fear of mistreatment, and other factors, PWID are far less likely to be vaccinated compared to other populations. In response, we propose to continue our collaboration with a prominent community based organization serving African American and Latino PWID. Our project will explore baseline hesitancy to vaccinate among PWID, identify barriers to vaccination, and then develop and evaluate messaging designed to increase COVID-19 vaccination among our target population of PWID through a clinical trial.

DETAILED DESCRIPTION:
People who inject drugs (PWID) experience disproportionate risk of being infected with SARS-CoV-2, the virus that causes COVID-19. Unfortunately, due to stigma, fear of mistreatment, and other factors, PWID are far less likely to be vaccinated compared to other populations. African American and Latino populations also face disproportionate risk of infection and far greater COVID-19 death rates compared to White populations, yet due to issues including longstanding medical mistrust are also far less likely to vaccinate. For African American and Latino PWID, COVID-related risks increase even further and vaccination becomes even more unlikely.

In response, we propose to continue our collaboration with New York Harm Reduction Educators (NYHRE) a prominent New York City community based organization serving African American and Latino PWID. To increase SARS-CoV-2 vaccination among our target population, we will first assemble a community advisory board (CAB) that we will consult at all phases of the project.

Next, we will recruit a separate sample of PWID (n=500) via respondent driven sampling to evaluate intervention materials as part of a clinical trial. Upon enrollment, participants will be offered a free vaccination against SARS-CoV-2. Those who do not initially vaccinate will be randomized into one of two intervention groups: a no video group, and a video text group. The no video group will receive weekly text messages designed to address barriers to vaccination identified in formative research. The video text group will receive the same texts, along with links to videos we develop with NYHRE staff and clients to address barriers to SARS-CoV-2 vaccination. Our intervention will track response rates in both groups. Primary outcome measures will be vaccination within the initial weeks following enrollment and the subsequent intervention period by treatment group. Additional outcomes will include vaccination rates by demographic, including race/ethnicity and primary language (i.e. do English speaking participants respond differently to specific intervention components compared to monolingual Spanish speakers).

If shown successful this approach can be replicated with additional populations that experience health disparities, and in different languages across the United States.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be age 18 years or older, able to provide informed consent, able to read and understand English or Spanish. Participants must report injection drug use in the past 90 days. Participants also must not have previously vaccinated against SARS-CoV-2.

Exclusion Criteria:

* Pregnant women will be excluded. Likewise, adults unable to consent, individuals who are not yet adults (infants, children, teenagers) and prisoners will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 545 (Actual)
Dates: Start 2022-06-21 (Actual); Primary Completion 2025-11-25 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Vaccination uptake at baseline | baseline
  Did the participant vaccinate when offered?
Vaccination uptake at follow-up | up to 6 weeks
  Did the participant vaccinate when offered?
Vaccination series completion | up to 12 weeks
  Did the participant receive a second vaccine dose to complete the vaccination series?

SECONDARY OUTCOMES:
SARS-CoV-2 literacy at baseline | baseline
  Knowledge of COVID 19 as measured by correct responses to true/false questions.
SARS-CoV-2 literacy at follow-up | up to 12 weeks
  Knowledge of COVID 19 as measured by correct responses to true/false questions.
Secondary | baseline
  Attitudes toward vaccination and medical care at baseline
Secondary | up to 12 weeks
  Attitudes toward vaccination and medical care at follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- OnPoint NYC, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No